CLINICAL TRIAL: NCT04723329
Title: Lecturer at Cumhuriyet University
Brief Title: The Effect of Web-based Training on Gaining Exercise Behavior in Coronary Artery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Zeynep Unver, Principal Investigator, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Inonu University
Record Dates: First submitted 2021-01-13; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Decision Making; Exercise; Self Efficacy
Keywords: Exercise; web-based education; Patients
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- web-based education group (Experimental): Patients will be given a username and password to access the website. The change stage of the patients will be determined by the researcher with the Exercise Change Phase Short Question Form, and it will be ensured that they reach the educational content prepared according to the transtheoretic model. Motivating interviews will be provided to the patients to receive training on the website by contacting them one-on-one. In the following 1st and 3rd months, patients will be contacted individually again to confirm whether they follow the website, and they will be asked to fill in the scales on the website by providing consultancy on the issues they need. In the 6th month, the final test data will be obtained from the website using the same data collection forms.
  Interventions: Behavioral: Web-based exercise training based on the transtheoretic model
- Control Group (No Intervention): In the first interview, the patients in the control group will be collected data and contact information will be obtained using the Patient Information Form, Exercise Change Phase Short Question Form, Change Processes Scale, Decision Making Balance Scale and Self-Efficacy Scale. Later, patients will be given their username and password so that they can log into the website where the scales are located in order to apply the final test. No intervention will be applied to the patients in the control group. At the end of the 6th month, the same scales will be applied on the website as a final test. At the end of the study, it is aimed to gain exercise behavior to the patients in the control group.

INTERVENTIONS:
Behavioral: Web-based exercise training based on the transtheoretic model — Motivating interviews will be provided to the patients to receive training on the website by contacting them one-on-one. In the following 1st and 3rd months, patients will be contacted individually again to confirm whether they follow the website, and they will be asked to fill in the scales on the website by providing consultancy on the issues they need. In the 6th month, the final test data will be obtained from the website using the same data collection forms.
  Arms: web-based education group

SUMMARY:
The aim of this thesis is; The aim of this study is to examine the effect of web-based training based on transtheoretic model on exercise behavior in patients with coronary artery disease.

The research is a randomized controlled trial. 114 patient who meet the conditions for research will be included in the study. In collecting data, the Patient Information Form, Exercise Change Phase Short Question Form, Exercise Change Processes Scale, Exercise Decision Making Scale and Exercise Self-Efficacy Scale developed by the researcher will be used.

DETAILED DESCRIPTION:
In the first interview, the patients in the experimental group will be collected data and contact information will be obtained using the Patient Information Form, Exercise Change Phase Short Question Form, Exercise Change Processes Scale, Exercise Decision Making Balance Scale and Exercise Self-Efficacy Scale as a pre-test. Then, the patients will be given their username and password to log into the website. The change stage of the patients will be determined by the researcher with the Exercise Change Phase Short Question Form, and it will be ensured that they reach the educational content prepared according to the transtheoretic model. Motivating interviews will be provided for the patients to receive training on the website by contacting them one-on-one. In the following 1st and 3rd months, the patients will be contacted individually again to confirm whether they follow the website, and they will be asked to fill the scales on the website by providing consultancy on the issues they need. In the 6th month, the final test data will be obtained from the website using the same data collection forms.

The patients in the control group will be collected data and contact information will be obtained at the first interview using the Patient Information Form, Exercise Change Phase Short Question Form, Change Processes Scale, Decision Making Balance Scale and Self-Efficacy Scale. Later, patients will be given their username and password so that they can log into the website where the scales are located in order to apply the final test. No intervention will be applied to the patients in the control group. At the end of the 6th month, the same scales will be applied on the website as a final test. At the end of the study, the patients in the control group will be able to access the exercise training content prepared for the purpose of gaining exercise behavior on the website.

Nursing Initiative The patients in the experimental group will be given a web-based exercise training based on the transtheoretic model according to the stages of change they are in.

Interference Material As the initiative material, the participants; A website will be established where they can log in with an individually given username and password. As the content; The harms of sedentary life, the benefits of exercise on general health, especially its effects on reducing heart diseases and risks, and materials for gaining exercise behavior will be included.

ELIGIBILITY:
Inclusion Criteria:

* Being literate
* Having internet access and using it comfortably, Independent in daily life activities

Exclusion Criteria:

* Have any physical and psychological problems that prevent exercising
* Those who do not intend to exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Exercise Change Stage | up to 6 months
  Exercise Change Stage Short Question Form is an 5 item scale. 1=Exercising regularly for more than 6 months, 2=Exercising regularly for less than 6 months, 3=Does not exercise but intends to do it within 30 days, 4=Does not exercising but intends to start within 6 months, 5=Does not exercise and does not intend to start within 6 months
Exercise Change Processes Scale | up to 6 months
  Change Processes Scale is an 28 item scale.Individuals in the scale do not agree with each statement using a 5-point Likert scale. is determined. Each individual in scale how much to exercise in the condition stated in item he often does a It is determined by the grading score. From the interviewee, the items of this scale by reading "1 = never" for each item, "2 = rarely", "3 = occasionally", "4 = often", "5 very often" the most suitable for him He is asked to select and mark the one. Scale, item points of all subscales score obtained from averages It is evaluated according to the average.There are cognitive and behavioral processes that facilitate change in the Exercise Change Processes Scale. The overall Cronbach's alpha coefficient of the scale is 0.95, and it was determined as 0.91 for cognitive processes with sub-dimensions and 0.93 for behavioral processes.
Exercise Decision-Making Balance | up to 6 months
  Change Processes Scale is an 10 item scale. Total score of the scale, the perceived benefit of exercising is total of the total score of perceived damage It is obtained by subtraction. Your result negative (-), in decision-making balance the perceived harms of exercise dominant, positive (+), decision exercising in a giving balance a sign that the perceived benefits are dominant does. The highest score that can be obtained from the scale 25 is the lowest score is 5.
Exercise Self-Efficacy Scale | up to 6 months
  Self-Efficacy Scale is an 6 item scale.From scale the highest score an individual can get is 30, low score is 6. In the evaluation of the scale; The higher the item score average, the higher the individual's selfishness.

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep UNVER, Malatya, Turkey (Türkiye)